CLINICAL TRIAL: NCT02618161
Title: A Randomised Feasibility Trial to Investigate the Timing of HDR Brachytherapy With EBRT in Intermediate and High Risk Localised Prostate CAncer Patients and Its Effects on Toxicity and Quality of Life
Brief Title: Timing of HDR With EBRT in Localised Prostate Cancer,Toxicity and Quality of Life Assessment
Acronym: THEPCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0845
Record Dates: First submitted 2015-10-08; First posted 2015-12-01 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
Keywords: EBRT and HDR Brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): HDR Brachytherapy single dose of 15 Gy followed by EBRT of 46 Gy in 23 fractions and Androgen deprivation therapy 6 months to 3 years, (sequencing of HDR followed by EBRT)
  Interventions: Radiation: HDR Brachytherapy; Radiation: External beam Radiotherapy
- ARM B (Active Comparator): External Beam Radiotherapy (EBRT) of 46 Gy in 23 fractions, followed by single dose of HDR brachytherapy of 15 Gy boost and Androgen deprivation therapy 6 months to 3 years (timing of HDR Brachytherapy Treatment is changed compared to ARM A)
  Interventions: Radiation: HDR Brachytherapy; Radiation: External beam Radiotherapy

INTERVENTIONS:
Radiation: HDR Brachytherapy — HDR Brachytherapy, a single dose of 15 Gy delivered to prostate
Radiation: External beam Radiotherapy — External beam Radiotherapy, a dose of 46 Gy in 23 fractions delivered to prostate

SUMMARY:
TITLE Timing of HDR brachytherapy with EBRT in intermediate and high risk localised Prostate CAncer patients and its effects on Toxicity and Quality of life - randomised feasibility trial.

SHORT TITLE THEPCA trial Protocol Version Number and Date Version 2.1, dated 16 DEC 2014 Study Duration Recruitment Duration 18-24 months

Study Centre Southend University Hospital NHS Foundation Trust

Objectives Assessment of acute toxicities: Genitourinary, gastrointestinal and sexual dysfunction at various time points.

Number of Participants 50 participants

Main Inclusion Criteria

* Patient age >18 years
* Histologically diagnosed Prostate cancer, stages T1b-T3bN0M0
* Any Gleason score
* Any PSA level
* Patient able to consent and fill in the questionnaires Exclusion Criteria - Previous TURP/HoLEP Laser Prostatectomy
* Any Metastatic Disease
* IPSS>20
* Pubic arch interference
* Lithotomy position or anaesthesia not possible
* Rectal fistula
* Prior pelvic radiotherapy Statistical Methodology and Analysis Percentages of adverse events will be compared using Fisher's Exact Test. Toxicity score means will be compared using two-sample permutation t-tests, and PSA relapse-free survival will be estimated using Kaplan-Meier and compared using log-rank tests.

DETAILED DESCRIPTION:
The role of radiotherapy in management of prostate cancer significantly changed over the last few decades with the developments in Brachytherapy, External Beam Radiotherapy (EBRT), Intensity modulated Radiotherapy (IMRT) and Image guided Radiotherapy (IGRT). One of the challenging factors of Radiotherapy treatment of localised prostate cancer is acute and late Genitourinary and Gastrointestinal toxicities. There are several studies and case series published in literature assessing the toxicities developed during EBRT and Brachytherapy treatment for prostate cancer EBRT and Brachytherapy emerged as the main stay of localised prostate cancer treatment in recent years. The low risk localised prostate cancers can be treated with low dose brachytherapy or by prostatectomy, whereas the intermediate and high risk localised prostate cancers are usually treated with EBRT alone or along with HDR brachytherapy. The recent European guidelines suggest that there is no consensus regarding the timing of HDR brachytherapy and EBRT. The schedules vary in different institutions where HDR boost can be given either before or after EBRT. Few centres deliver HDR in-between the fractions of EBRT.

The EBRT doses range from 37.5Gy in 15 fractions to 45Gy in 25 fractions when given with HDR. The total HDR brachytherapy dose can be delivered in fractions, however a single dose of 15Gy is gaining acceptance across the world due to its logistical advantage. The Time gap between the two Radiotherapy modes of delivery is generally within 21 days.

There is no consensus about the timing of HDR brachytherapy (BT) when treated along with EBRT. The advantages of using HDR Brachytherapy before EBRT are that the investigators could potentially identify patients who are not suitable for brachytherapy early in the treatment process. It is essential to know whether there is any significant difference in toxicities and treatment outcome especially acute urinary toxicity amongst the two treatment approaches. It will be done by a simple 1:1 ratio randomisation which will only be possible if a participant meets the inclusion and exclusion criteria.

Brachytherapy procedure Procedure will be carried out at the surgical theatres in Southend University Hospital.

1. Patients will undergo prostate implantation under general or spinal anesthetic using a Transrectal ultrasound guided transperineal technique.
2. Imaging according to local practice using ultrasound, CT and or MR will be undertaken
3. The CTVp is defined by the prostate capsule and extended to include any extra capsular or seminal vesicle disease. A volumetric expansion of 3mm constrained to the rectum posteriorly is then added. This defines the PTV.
4. Catheter reconstruction and dwell time definition is then undertaken to provide a treatment plan for approval by the treating clinician.
5. Treatment is delivered once an optimized plan has been approved
6. After completion of treatment in the brachytherapy room the implant catheters and urinary catheter are removed; no anesthesia is required for this procedure.
7. The patient will return to the ward and may be discharged home later the same day or the following day Dose prescription A dose of 15Gy in a single treatment exposure defined at the 100% isodose which is the minimum tumour isodose to cover the PTV.

PTV recommendations D90: ≥15Gy V100: ≥95%

Organs at risk tolerance doses:

Rectum D2cc 12Gy Rectum V100 <15Gy Urethra D10 <17.5Gy Urethra D30 <16.5Gy Urethra V150 0cc

External Beam Radiation Therapy (EBRT) EBRT would be given to prostate and seminal vesicles only, using either Intensity Modulated Radiotherapy (IMRT) or Volumetric Arc radiotherapy (VMAT) to a dose of 4600cGy in 23 fractions over four and half weeks. The Dose Volume Histogram (DVH) would be according to the local radiotherapy protocol. The gap between BT and EBRT irrespective of their sequence should not exceed more than 3 weeks. Therefore the total Radiotherapy treatment time should be up to seven and half weeks Patients will receive neo-adjuvant and adjuvant anti androgen therapy between 6 months to 3 years according to the risk stratification of the disease as per standard of care All statistical significance testing will be at the 5% significance level. For the IPSS and IIEFS scale scores, the two means at each of the follow-up assessments will be compared using a two-sided permutation t-test using 1000000 random permutations, and the 95% confidence limits for the difference between the means will be calculated using a bootstrap using 9999 re-samplings. There will also be an assessment of trends in the scores through time using a repeated measures analysis of variance on the four follow-up scores with the baseline score as a covariate. For categorical data based on adverse events percentages will be compared using Fisher's Exact Test. In this small study it will be possible to carry out the full combinatorial calculations for Fisher's Exact Test (whereas in a main study 10000 random permutations will be obtained in a Monte Carlo approach.) For differences between percentages the 95% confidence limits will be obtained using Newcombe's Hybrid Score Interval method. For the secondary analysis Prostate-specific antigen relapse-free survival using the Kaplan-Meier method, with a test for difference between the survival curves using the log-rank test with the P-value obtained using permutation test with 10000 permutations. Cox proportional hazards multiple regression will also be used to assess the effects of covariates on survival, with model comparisons carried out using likelihood ratio tests. The analyses will be performed using the computer program R. All randomised participants will be included in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years
* Histologically diagnosed Prostate cancer, stages T1b-T3bN0M0
* Any Gleason score
* Any PSA level
* Patient able to consent and fill in the questionnaires

Exclusion Criteria:

* Previous TURP/HoLEP Laser Prostatectomy
* Any Metastatic Disease
* IPSS>20
* Pubic arch interference
* Lithotomy position
* If Anaesthesia is not possible
* Rectal fistula
* Prior pelvic radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Prospective assessment of genitourinary toxicities according to the treatment sequence of HDR Brachytherapy and EBRT | 12 months
  The Genitourinary toxicities are assessed according to CTCAE grading of toxicities (especially grade 3 and 4)

SECONDARY OUTCOMES:
Biochemical response and survival | 12 months
  PSA response in ug/L and its relation to survival rates at the end of year 1 follow up
Gastrointestinal toxicities according to the treatment sequence of HDR Brachytherapy and EBRT | 12 months
  Assessment of all CTCAE v4.0 grades of GI toxicities in both arms and the difference if any arise.
Radiotherapy Planning Challenges including Image Guided Radiotherapy | 12 months
  Assessment of timescales in planning the Radiotherapy and Brachytherapy once the patients entered in the trial and the number of patients received IGRT in the both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Imtiaz Ahmed, MRCP FRCR, Principal Investigator — Southend University Hospital NHS Foundation Trust
Locations (1):
- Southend Hospital, Westcliff-on-Sea, Essex, United Kingdom